CLINICAL TRIAL: NCT01117350
Title: A 24-week, Multicenter, International, Randomized (1:1), Parallel-group, Open-label, Comparative Study of Insulin Glargine Versus Liraglutide in Insulin-naïve Patients With Type 2 Diabetes Treated With Oral Agents and Not Adequately Controlled, Followed by a 24-week Extension Period With Insulin Glargine for Patients Not Adequately Controlled With Liraglutide
Brief Title: Efficacy Assessment of Insulin Glargine Versus LiraglutidE After Oral Agents Failure
Acronym: EAGLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_C_03680; 2010-018437-21 (EudraCT Number); U1111-1116-9684 (Other: UTN)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Liraglutide; Metformin

ARMS (2):
- Insulin Glargine (Experimental): Insulin glargine administered once a day, in the morning or in the evening, at the most convenient time. The time of injection, once chosen was to remain unchanged during the whole duration of the study.
  The starting dose was 0.2 Unit per kilogram of body weight or 10 Units. Patients were empowered to adjust their insulin doses, under strict investigator's supervision. Insulin titration (by 2 or 4 Units) was done every 3 days according to the median value of Fasting Plasma Glucose (FPG) of the last 3 days. The goal was to achieve 70 < FPG ≤ 100 mg/dL (3.9 < FPG ≤ 5.5 mmol/L). Minor deviations from the titration scheme could be allowed, based on Investigator's judgment and patient's situation.
  Interventions: Drug: Insulin glargine; Drug: Metformin
- Liraglutide (Active Comparator): Liraglutide administered once a day, in the morning or in the evening, at the most convenient time. The time of injection , once chosen was to remain unchanged during the whole duration of the study.
  The dose was 0.6 mg/day during the first week, 1.2 mg/day during the second week and 1.8 mg/day until week 24. The dose might be decreased to 1.2 mg for safety reasons (e.g. gastro-intestinal tolerability), based on Investigator's judgment.
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: Insulin glargine — 100 Units/mL solution for injection in a pre-filled SoloStar pen
  Other Names: Lantus®
  Arms: Insulin Glargine
Drug: Liraglutide — 6 mg/mL solution for injection in a 3-mL pre-filled pen (18mg)
  Other Names: Victoza®
  Arms: Liraglutide
Drug: Metformin — Metformin was a background treatment, mandatory for each patient randomized in the study (at the minimum dose of 1g/day). It was not supplied by the sponsor.

SUMMARY:
Primary objective:

To demonstrate the superiority of insulin glargine over liraglutide in terms of percentage of patients reaching a Glycosylated Haemoglobin (HbA1c) < 7% at the end of the comparative period (24 weeks) in Type 2 diabetic patients failing lifestyle management and oral agents

Secondary objectives of the comparative period (24 weeks):

>To assess the effect of insulin glargine in comparison with liraglutide on:

* HbA1c level
* Percentage of patients whose HbA1c has decreased but remains >= 7% at the end of the comparative period
* Percentage of patients whose HbA1c has increased at the end of the comparative period
* Fasting Plasma Glucose (FPG)
* 7-point Plasma Glucose (PG) profiles
* Hypoglycemia occurrence
* Body weight
* Adverse events

Objectives of the extension period (24 weeks):

>To assess the effect of insulin glargine in patients not adequately controlled with liraglutide on:

* HbA1c level
* FPG
* 7-point PG profiles
* Hypoglycemia occurrence
* Body weight
* Adverse events

DETAILED DESCRIPTION:
Maximum estimated study duration per patient: either 27 weeks (patients randomized to insulin glargine arm) or 51 weeks (patients randomized to liraglutide arm) broken down as follow:

* A 2-week of screening period,
* A 24-week comparative period,
* A 24-week extension period (only for patients treated with liraglutide, not adequately controlled at the end of the comparative period),
* A 1-week follow-up period

ELIGIBILITY:
Inclusion criteria (comparative period):

* Patients With Type 2 Diabetes diagnosed for at least 1 year,
* Treated with lifestyle interventions and metformin at the maximum tolerated dosage (with a minimum daily dosage of 1g), either alone or in combination with an oral insulin secretagogue (sulfonylurea, glinide or DiPeptidyl Peptidase IV inhibitor), for more than 3 months,
* 7.5% < HbA1c <= 12%,
* Body Mass Index (BMI) between 25 and 40 kg/m2 inclusively,
* Ability and willingness to perform PG (Plasma Glucose) self monitoring using the sponsor-provided glucose meter and to complete the patient diary,
* Willingness and ability to comply with the study protocol,
* Signed informed consent obtained prior to any study procedure.

Inclusion criteria (extension period):

* Patients treated with liraglutide (at the maximal tolerated dosage), having a mean FPG ≥ 250 mg/dL at visit 10 (Week 12) or visit 11 (Week 18), or a HbA1c≥ 7% at visit 12 (Week 24)
* Dosage of metformin compliant with the inclusion criteria of visit 1 (i.e. maximum tolerated dosage, with a minimum daily dosage of 1g), and maintained stable during the comparative period.

Exclusion criteria:

* Previous treatment with Glucagon Like Peptide-1 analogues or insulin in the past year (except in case of temporary treatment for gestational diabetes, surgery, hospitalization...),
* Treatment with thiazolidinediones or α-Glucosidases inhibitors within 3 months prior to study entry,
* Diabetes other than Type 2 diabetes (e.g. secondary to pancreatic disorders, drug or chemical agents intake),
* Pregnant women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraceptive method),
* Lactating women,
* Hospitalized patients (except hospitalization for routine diabetes check-up),
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to study entry, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study, documented by a retina examination within 2 years prior to study entry,
* Impaired renal function (creatinine clearance < 60 mL/mn),
* Impaired hepatic function (Alanine Aminotransferase, Aspartate Aminotransferase 2.5 times the upper limit of normal range),
* Personal or family history of medullary thyroid carcinoma,
* Multiple endocrine neoplasia syndrome type 2,
* Severe gastro-intestinal disease (including inflammatory bowel disease or diabetic gastroparesis),
* Congestive heart failure,
* History of acute pancreatitis,
* Treatment with corticosteroids with potential systemic action for more than 10 days within 3 months prior to study entry,
* Alcohol or drug abuse in the past 5 years,
* History of sensitivity to the study drugs or to drugs with a similar chemical structure.
* Night shift worker,
* Presence of any condition (medical, psychological, social or geographical), current or anticipated that would compromise the patients safety or limit the patient successful participation in the study,
* Participation in a clinical trial (drug or device) within 3 months prior to study entry,
* Refusal or inability to give informed consent to participate in the study,
* Patient is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

Additional exclusion criteria for the extension period:

* Treatment with oral antidiabetic drugs other than metformin and patient's usual sulfonylurea if any, or with insulin during the comparative period (except in case of an emergency, for a period of time less than 7 days),
* Treatment with corticosteroids with potential systemic action within the last 3 months of the comparative period.
* History of sensitivity to insulin glargine.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 978 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (136):
- United States (45):
  - Investigational Site Number 840023, Birmingham, Alabama
  - Investigational Site Number 840002, Goodyear, Arizona
  - Investigational Site Number 840047, Phoenix, Arizona
  - Investigational Site Number 840017, La Jolla, California
  - Investigational Site Number 840036, La Mesa, California
  - Investigational Site Number 840037, Loma Linda, California
  - Investigational Site Number 840045, Long Beach, California
  - Investigational Site Number 840048, Mission Hills, California
  - Investigational Site Number 840033, Mission Viejo, California
  - Investigational Site Number 840019, Palm Springs, California
  - Investigational Site Number 840039, San Diego, California
  - Investigational Site Number 840042, San Diego, California
  - Investigational Site Number 840043, Tustin, California
  - Investigational Site Number 840028, Denver, Colorado
  - Investigational Site Number 840034, Grand Junction, Colorado
  - Investigational Site Number 840026, Longmont, Colorado
  - Investigational Site Number 840022, Lawrenceville, Georgia
  - Investigational Site Number 840029, Roswell, Georgia
  - Investigational Site Number 840009, Arlington Heights, Illinois
  - Investigational Site Number 840051, Springfield, Illinois
  - Investigational Site Number 840050, Indianapolis, Indiana
  - Investigational Site Number 840031, Kansas City, Kansas
  - Investigational Site Number 840004, Paducah, Kentucky
  - Investigational Site Number 840010, Rockville, Maryland
  - Investigational Site Number 840038, Eagan, Minnesota
  - Investigational Site Number 840030, Minneapolis, Minnesota
  - Investigational Site Number 840012, St Louis, Missouri
  - Investigational Site Number 840044, St Louis, Missouri
  - Investigational Site Number 840015, Atco, New Jersey
  - Investigational Site Number 840008, Blackwood, New Jersey
  - Investigational Site Number 840027, Mineola, New York
  - Investigational Site Number 840011, Staten Island, New York
  - Investigational Site Number 840005, Hickory, North Carolina
  - Investigational Site Number 840052, Winston-Salem, North Carolina
  - Investigational Site Number 840049, Fargo, North Dakota
  - Investigational Site Number 840006, Bryan, Ohio
  - Investigational Site Number 840035, Cincinnati, Ohio
  - Investigational Site Number 840016, Carnegie, Pennsylvania
  - Investigational Site Number 840020, Uniontown, Pennsylvania
  - Investigational Site Number 840024, Rapid City, South Dakota
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840007, Dallas, Texas
  - Investigational Site Number 840013, Houston, Texas
  - Investigational Site Number 840014, Renton, Washington
  - Investigational Site Number 840046, Spokane, Washington
- Austria (7):
  - Investigational Site Number 040-006, Salzburg
  - Investigational Site Number 040-007, Salzburg
  - Investigational Site Number 040-003, Stockerau
  - Investigational Site Number 040-005, Vienna
  - Investigational Site Number 040-002, Vienna
  - Investigational Site Number 040-001, Vienna
  - Investigational Site Number 040-004, Vienna
- Brazil (6):
  - Investigational Site Number 076-004, Belém
  - Investigational Site Number 076-007, Fortaleza
  - Investigational Site Number 076-001, Fortaleza
  - Investigational Site Number 076-006, Fortaleza
  - Investigational Site Number 076-005, Marília
  - Investigational Site Number 076-002, São Paulo
- Canada (6):
  - Investigational Site Number 124-003, Mississauga
  - Investigational Site Number 124-001, Montreal
  - Investigational Site Number 124-006, Montreal
  - Investigational Site Number 124-004, Toronto
  - Investigational Site Number 124-008, Vancouver
  - Investigational Site Number 124-007, Victoria
- Czechia (5):
  - Investigational Site Number 203001, Hradec Králové
  - Investigational Site Number 203003, Krnov
  - Investigational Site Number 203005, Kroměříž
  - Investigational Site Number 203002, Olomouc
  - Investigational Site Number 203006, Prague
- Finland (4):
  - Investigational Site Number 246003, Harjavalta
  - Investigational Site Number 246001, Kuopio
  - Investigational Site Number 246002, Oulu
  - Investigational Site Number 246004, Turku
- France (14):
  - Investigational Site Number 250-007, Annecy
  - Investigational Site Number 250-017, Bois-Guillaume
  - Investigational Site Number 250-003, Boulogne-Billancourt
  - Investigational Site Number 250-011, Brest
  - Investigational Site Number 250-008, Cahors
  - Investigational Site Number 250-012, Corbeil-Essonnes
  - Investigational Site Number 250-009, La Rochelle
  - Investigational Site Number 250-004, Le Creusot
  - Investigational Site Number 250-006, Mantes-la-Jolie
  - Investigational Site Number 250-021, Nanterre
  - Investigational Site Number 250022, Strasbourg
  - Investigational Site Number 250-020, Strasbourg
  - Investigational Site Number 250-002, Toulouse
  - Investigational Site Number 250-016, Vénissieux
- Greece (3):
  - Investigational Site Number 300003, Athens
  - Investigational Site Number 300004, Athens
  - Investigational Site Number 300001, Haidari, Athens
- Investigational Site Number 372001, Dublin, Ireland
- Israel (3):
  - Investigational Site Number 376004, Hadera
  - Investigational Site Number 376002, Petah Tikva
  - Investigational Site Number 376003, Tel Aviv
- Mexico (4):
  - Investigational Site Number 484004, Guadalajara
  - Investigational Site Number 484001, México
  - Investigational Site Number 484002, México
  - Investigational Site Number 484003, Zapopan
- Netherlands (7):
  - Investigational Site Number 528004, 's-Hertogenbosch
  - Investigational Site Number 528001, Beek
  - Investigational Site Number 528006, Enschede
  - Investigational Site Number 528002, Hoogeveen
  - Investigational Site Number 528007, Nijverdal
  - Investigational Site Number 528003, Rotterdam
  - Investigational Site Number 528005, Woerden
- Russia (8):
  - Investigational Site Number 643-009, Kazan'
  - Investigational Site Number 643008, Kirov
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643004, Saint Petersburg
  - Investigational Site Number 643006, Samara
  - Investigational Site Number 643007, Samara
  - Investigational Site Number 643005, Saratov
  - Investigational Site Number 643003, St-Ptetersburg
- Slovakia (5):
  - Investigational Site Number 703002, Bratislava
  - Investigational Site Number 703004, Košice
  - Investigational Site Number 703001, Nitra
  - Investigational Site Number 703005, Nové Mesto nad Váhom
  - Investigational Site Number 703003, Žilina
- Spain (10):
  - Investigational Site Number 724007, Bilbao
  - Investigational Site Number 724006, Cadiz
  - Investigational Site Number 724001, Las Palmas de Gran Canaria
  - Investigational Site Number 724005, Lleida
  - Investigational Site Number 724008, Madrid
  - Investigational Site Number 724003, Málaga
  - Investigational Site Number 724009, Sabadell
  - Investigational Site Number 721002, Valencia
  - Investigational Site Number 724004, Valencia
  - Investigational Site Number 724010, Vigo
- Sweden (6):
  - Investigational Site Number 752-03, Ängelholm
  - Investigational Site Number 752-002, Gothenburg
  - Investigational Site Number 752-005, Karlskoga
  - Investigational Site Number 752-006, Motala
  - Investigational Site Number 752-007, Örebro
  - Investigational Site Number 752-001, Stockholm
- Turkey (Türkiye) (2):
  - Investigational Site Number 792-001, Antalya
  - Investigational Site Number 792-002, Istanbul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on July 23, 2010. The 24-week comparative period was completed on October 5, 2012.
  The extension period was initiated on March 24, 2011 and completed on March 6, 2013.
Pre-assignment Details: A total of 1456 patients were screened in 136 centers, in 17 countries (Austria, Brazil, Canada, Czech Republic, Finland, France, Greece, Ireland, Israel, Mexico, Netherlands, Russian Federation Slovakia, Spain, Sweden, Turkey, USA). Among them, 478 (32.8%) patients were not randomized (main reason was Glycosylated Haemoglobin A1c out of range).
Groups:
- Insulin Glargine: Insulin glargine starting dose: 0.2 Unit per kilogram of body weight or 10 Units. Insulin titration (by 2 or 4 Units) every 3 days according to the median value of Fast Plasma Glucose of the last 3 days
- Liraglutide (Comparative Period)/ Insulin Glargine (Extension): Liraglutide dose: 0.6 mg/day during the first week, 1.2 mg/day during the second week and 1.8 mg/day until week 24 (comparative period)
  For patients included in the extension period: Insulin Glargine (dosing same as above)
Period: Comparative Period
Arm/Group | Insulin Glargine | Liraglutide (Comparative Period)/ Insulin Glargine (Extension)
Started | 489 (STARTED: randomized) | 489
TREATED = Safety Population | 484 (Safety population: all randomized and treated patients (received at least one dose)) | 481
mITT Population | 474 (modified Intent-To-Treat population: treated patients with at least one efficacy post-baseline value) | 470
Completed | 447 | 414
Not Completed | 42 | 75
Not completed — Not Treated | 5 | 8
Not completed — Adverse Event | 6 | 33
Not completed — Lost to Follow-up | 11 | 7
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Protocol Violation | 8 | 12
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Move to another city/country | 2 | 1
Period: Extension Period
Arm/Group | Insulin Glargine | Liraglutide (Comparative Period)/ Insulin Glargine (Extension)
Started | 0 | 210 (STARTED: patients having completed the comparative period and eligible for the extension period)
TREATED = Safety Population (Extension) | 0 | 160 (Safety population (extension): treated with insulin glargine during the extension period)
mITT Population (Extension) | 0 | 154 (mITT (extension): treated patients with at least 1 efficacy value both at entry and during extension)
Completed | 0 | 147
Not Completed | 0 | 63
Not completed — Not included in extension, not treated | 0 | 50
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Inclusion criteria not respected | 0 | 1
Not completed — Prohibited medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified-Intent-to-treat (mITT) population: all patients who were randomized, received at least one dose of Interventional Product (IP), and had at least one post-baseline assessment during comparative period of any primary or secondary efficacy variables
Groups:
- Liraglutide: Liraglutide dose: 0.6 mg/day during the first week, 1.2 mg/day during the second week and 1.8 mg/day until week 24.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | Liraglutide | Total
Number analyzed (Participants) | 474 | 470 | 944
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.07 (8.78) | 57.44 (8.85) | 57.25 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 207 | 431
  Male | 250 | 263 | 513
Body Mass Index (BMI) at week -2 [Mean (Standard Deviation); unit: kg/m²] | 32.00 (4.24) | 31.75 (4.12) | 31.88 (4.18)
Duration of Type 2 diabetes [Median (Inter-Quartile Range); unit: years] | 8.54 [5.20 to 12.38] | 8.41 [4.80 to 11.69] | 8.49 [4.94 to 12.17]
At least one diabetic late complication [Number; unit: participants] — Diabetic late complications: myocardial infarction, angina pectoris, coronary artery disease, heart failure, stroke, transient ischemic attack, peripheral vascular disease, diabetic neuropathy, diabetic nephropathy, diabetic retinopathy
  participants
    Yes | 212 | 223 | 435
    No | 262 | 247 | 509
Glycosylated Hemoglobin A1c (HbA1c) at week -2 [Mean (Standard Deviation); unit: percent] | 9.04 (1.10) | 9.11 (1.09) | 9.07 (1.09)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Whose Glycosylated Haemoglobin (HbA1c) <7% at the End of the Comparative Period
Description: The value at the end of the comparative period was defined as the last available HbA1c value measured during the comparative period plus 14 days after the last dose of Investigational Product (i.e. last-observation-carried-forward [LOCF] value).
Time Frame: week 12, week 24
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had at least one HbA1c value on treatment during the comparative period.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 467 | 458
percentage of participants | 48.4 | 45.9
Statistical Analysis 1: Comparison: Insulin Glargine vs Liraglutide; Superiority testing H0: Rate measured with insulin glargine = rate measured with liraglutide H1: Rate measured with insulin glargine ≠ rate measured with liraglutide Sample size calculation (465 randomized patients per arm) was based on the assumption of an expected success rate of 46% with insulin glargine and 35% with liraglutide, an alpha risk of 5% (2-sided) and a power of 90%, taking into account an estimated non evaluability rate of 10%; Test type: Superiority or Other; p = 0.439, Chi-squared — If superiority not demonstrated, switching from superiority to non-inferiority considered. Conclusion of non-inferiority reached if lower limit of 2-sided 95% confidence interval of the difference (insulin glargine - liraglutide) > or = to - 3.5%; Mean Difference (Final Values) = 2.54, 95% CI 2-sided [-3.88 to 8.93]

2. Secondary Outcome: Percentage of Patients Whose Glycosylated Haemoglobin (HbA1c) Has Decreased But Remains ≥7% at the End of the Comparative Period
Description: Percentage of patients with:
  * HbA1c value at end of the comparative period (LOCF) lower than HbA1c baseline value
  AND
  * HbA1c value at end of the comparative period (LOCF) ≥7%
Time Frame: baseline (week -2), week 12, week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 467 | 458
percentage of participants | 47.1 | 46.3

3. Secondary Outcome: Percentage of Patients Whose Glycosylated Haemoglobin (HbA1c) Has Increased at the End of the Comparative Period
Description: Percentage of patients with HbA1c value at end of the comparative period (LOCF) higher than HbA1c baseline value
Time Frame: baseline (week -2), week 12, week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 467 | 458
percentage of participants | 4.1 | 6.6

4. Secondary Outcome: Glycosylated Haemoglobin (HbA1c): Change From Baseline to the End of Comparative Period
Description: Change in HbA1C from baseline to the last observation carried forward (LOCF) measured during the comparative period = LOCF value - baseline value
Time Frame: baseline (week -2), week 12, week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 467 | 458
percent | -1.92 (1.22) | -1.81 (1.33)

5. Secondary Outcome: Glycosylated Haemoglobin (HbA1c): Change From Beginning to the End of the Extension Period
Description: Change in HbA1C from beginning of the extension period (week 24) to the last observation carried forward (LOCF) measured during the extension period = LOCF value - week 24 value
Time Frame: week 24, week 36, week 48
Population: The population analyzed for this outcome measure consisted of the subset of mITT population (extension) who had HbA1c value both at beginning of the extension and at least one value on treatment during the extension period.
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Insulin Glargine (Extension Period): Insulin glargine starting dose: 0.2 Unit per kilogram of body weight or 10 Units. Insulin titration (by 2 or 4 Units) every 3 days according to the median value of Fast Plasma Glucose of the last 3 days
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 152
percent | -0.26 (1.11)

6. Secondary Outcome: Percentage of Patients Whose Glycosylated Haemoglobin (HbA1c) <7% at the End of the Extension Period
Description: Value at the end of the extension period defined as last available HbA1c value measured during the extension period (i.e. last observation carried forward (LOCF) value)
Time Frame: week 36, week 48
Population: The population analyzed for this outcome measure consisted of the mITT patients who had at least one HbA1c value on treatment during the extension period.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 154
percentage of participants | 22.7

7. Secondary Outcome: Self-Monitored Fasting Plasma Glucose (SMFPG) Measurements: Change From Baseline to the End of the Comparative Period
Description: SMFPG = mean value of Self-Monitored Fasting Plasma Glucose measurements over 3 consecutive days in the week before each visit
  Value at the end of the comparative period defined as last available value during the comparative period (i.e. last-observation-carried-forward [LOCF] value)
  Change = LOCF value - baseline value
Time Frame: baseline (week 0), week 6, week 12, week 18, week 24
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had at least one SMFPG value on treatment during the comparative period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 468 | 452
mg/dL | -65.25 (50.95) | -37.23 (47.31)

8. Secondary Outcome: Self-Monitored Fasting Plasma Glucose (SMFPG) Measurements: Change From Beginning to the End of the Extension Period
Description: SMFPG = mean value of Self-Monitored Fasting Plasma Glucose measurements over 3 consecutive days in the week before each visit
  Value at the end of the extension period defined as last available value during the extension period (i.e. last-observation-carried-forward [LOCF] value)
  Change = LOCF value - week 24 value
Time Frame: week 24, week 30, week 36, week 48
Population: The population analyzed for this outcome measure consisted of the subset of mITT (extension) patients who had SMFPG value both at beginning of the extension and at least one value on treatment during the extension period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 147
mg/dL | -44.63 (45.47)

9. Secondary Outcome: Self-Monitored 7-point Plasma Glucose (PG) Profile: Change From Baseline to the End of the Comparative Period
Description: Self-monitored 7-point plasma glucose profiles (before and 2 hours after the start of breakfast, lunch and dinner, and at bedtime) recorded on 3 consecutive days in the week before each visit
  Value at the end of the comparative period defined as last available value during the comparative period (i.e. last-observation-carried-forward [LOCF] value)
  Change = LOCF value - baseline value
Time Frame: baseline (week 0), week 12, week 24
Population: The population considered was the mITT population but due to missing values, different subsets of this mITT population were analyzed for each time point of the profile.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 474 | 470
mg/dL
  Before breakfast (N ig = 448 & N l = 409) | -65.92 (50.29) | -38.64 (46.17)
  After breakfast (N ig = 440 & N l = 397) | -66.70 (63.29) | -55.35 (61.56)
  Before lunch (N ig = 438 & N l = 404) | -50.16 (59.53) | -39.13 (58.78)
  After lunch (N ig = 433 & N l = 406) | -43.00 (58.42) | -41.82 (61.16)
  Before dinner (N ig = 434 & N l = 400) | -40.84 (58.88) | -36.88 (58.49)
  After dinner (N ig = 426 & N l = 396) | -42.6 (61.74) | -45.04 (60.42)
  At bedtime (N ig = 380 & N l = 351) | -43.11 (60.37) | -44.06 (59.80)

10. Secondary Outcome: Self-Monitored 7-point Plasma Glucose (PG) Profile: Change From Beginning to the End of the Extension Period
Description: Self-monitored 7-point plasma glucose profiles (before and 2 hours after the start of breakfast, lunch and dinner, and at bedtime) recorded on 3 consecutive days in the week before each visit
  Value at the end of the extension period defined as last available value during the extension period (i.e. last-observation-carried-forward [LOCF] value)
  Change = LOCF value - week 24 value
Time Frame: week 24, week 36, week 48
Population: The population considered was the mITT population (extension) but due to missing values, different subsets of this population were analyzed for each time point of the profile.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 154
mg/dL
  Before breakfast (N=143) | -46.13 (44.89)
  After breakfast (N=134) | -27.67 (52.37)
  Before lunch (N=131) | -20.32 (57.58)
  After lunch (N=134) | -11.50 (58.37)
  Before dinner (N=133) | -12.56 (54.57)
  After dinner (N=130) | -2.28 (54.55)
  At bedtime (N=127) | -14.94 (52.67)

11. Secondary Outcome: Body Weight: Change From Baseline to the End of the Comparative Period
Description: Change = Last weight value measured during the comparative period (LOCF value) - weight value at baseline
Time Frame: baseline (week 0), week 2, week 6, week 12, week 18, week 24
Population: The population analyzed for this outcome measure consisted of the subset of mITT patients who had at least one weight value on treatment during the comparative period.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 474 | 468
kg | 1.98 (3.95) | -2.99 (3.64)

12. Secondary Outcome: Body Weight: Change From Beginning to End of the Extension Period
Description: Change = Last weight value measured during the extension period (LOCF value) - weight value at beginning of the Extension Period (Week 24)
Time Frame: week 24, week 30, week 36, week 48
Population: The population analyzed for this outcome measure consisted of the mITT population (extension).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 154
kg | 4.35 (3.39)

13. Secondary Outcome: Daily Dose of Insulin Glargine
Time Frame: week 1, week 2, week 6, week 12, week 24
Population: The population considered was the mITT population but due to missing values, different subsets of this mITT population were analyzed at each week.
Measure: Mean (Standard Deviation); unit: Unit (U)
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 474
Unit (U)
  Start of treatment (N=472) | 13.39 (4.87)
  Week 1 (N=470) | 17.74 (6.52)
  Week 2 (N=470) | 22.06 (8.40)
  Week 6 (N=470) | 34.67 (17.03)
  Week 12 (N=463) | 44.40 (26.63)
  Week 18 (N=454) | 48.65 (31.03)
  Week 24 (N=459) | 51.67 (34.05)
  End comparative period (LOCF) (N=474) | 51.24 (33.93)

14. Secondary Outcome: Daily Dose of Liraglutide
Time Frame: week 1, week 2, week 6, week 12, week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Liraglutide
Number analyzed (Participants) | 470
mg
  Start of treatment (N=470) | 0.60 (0.00)
  Week 1 (N=463) | 0.91 (0.31)
  Week 2 (N=458) | 1.49 (0.33)
  Week 6 (N=444) | 1.72 (0.21)
  Week 12 (N=426) | 1.73 (0.19)
  Week 18 (N=415) | 1.74 (0.18)
  Week 24 (N=431) | 1.73 (0.21)
  End comparative period (LOCF) (N=470) | 1.71 (0.24)

15. Secondary Outcome: Daily Dose of Insulin Glargine Administered During the Extension Period
Time Frame: week 30, week 36, week 48
Population: The population considered was the mITT population (extension) but due to missing values, different subsets of this mITT population were analyzed at each week.
Measure: Mean (Standard Deviation); unit: Unit (U)
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 154
Unit (U)
  Start of treatment (N=154) | 15.77 (4.53)
  Week 30 (N=151) | 37.49 (15.70)
  Week 36 (N=150) | 46.21 (23.06)
  Week 48 (N=151) | 50.68 (27.33)

16. Secondary Outcome: Hypoglycemia Occurence: Number of Patients With at Least One Episode of Symptomatic / Severe Symptomatic Hypoglycemia During the Comparative Period
Description: Symptomatic hypoglycemia was defined as an event with clinical symptoms that were considered to result from hypoglycemia.
  Severe symptomatic hypoglycemia was defined as an event with clinical symptoms that were considered to result from hypoglycemia, requiring the assistance of another person for active administration of carbohydrate, glucagon or other countermeasure because the patient could not treat him/herself due to acute neurological impairment directly resulting from the hypoglycemia (assistance by another person when the patient could have treated him/herself was not considered as requiring assistance)and one of the following criteria:
  * The event was associated with a measured PG level < 36 mg/dL (2 mmol/L),
  * Or, in absence of PG value, the event was associated with neurological recovery attributable to the restoration of PG to normal, after oral carbohydrate, intravenous glucose or glucagon administration.
Time Frame: all across the comparative period (from week 0 to week 24)
Population: The population analyzed was the safety population i.e. all randomized and treated patients.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Liraglutide
Number analyzed (Participants) | 484 | 481
participants
  symptomatic hypoglycemia | 219 | 85
  severe symptomatic hypoglycemia | 0 | 2

17. Secondary Outcome: Hypoglycemia Occurence: Number of Patients With at Least One Episode of Symptomatic / Severe Symptomatic Hypoglycemia During the Extension Period
Description: as for outcome 16
Time Frame: all across the extension period (from week 24 to week 48)
Population: The population analyzed was the safety population (extension) i.e. all treated patients during the extension period.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine (Extension Period)
Number analyzed (Participants) | 160
participants
  symptomatic hypoglycemia | 58
  severe symptomatic hypoglycemia | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study from the time the patient signed the informed consent until 7 days after the last dose of study treatment.
Description: The population analyzed was the safety population defined for each of the 2 periods (comparative and extension) as the patients treated with at least one dose of the study treatment during the considered period.
Groups:
- Comparative Period: Insulin Glargine: Insulin glargine starting dose: 0.2 Unit per kilogram of body weight or 10 Units. Insulin titration (by 2 or 4 Units) every 3 days according to the median value of Fast Plasma Glucose of the last 3 days
- Comparative Period: Liraglutide: Liraglutide dose: 0.6 mg/day during the first week, 1.2 mg/day during the second week and 1.8 mg/day until week 24 (comparative period)
- Extension Period: Insulin Glargine: Following a treatment with liraglutide during the comparative period, those patients have received insulin glargine during the extension period.
  Insulin glargine starting dose: 0.2 Unit per kilogram of body weight or 10 Units. Insulin titration (by 2 or 4 Units) every 3 days according to the median value of Fast Plasma Glucose of the last 3 days
Arm/Group | Comparative Period: Insulin Glargine | Comparative Period: Liraglutide | Extension Period: Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 11/484 | 15/481 | 5/160
Other Adverse Events (participants affected / at risk) | 92/484 | 239/481 | 22/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Comparative Period: Insulin Glargine (N=484) | Comparative Period: Liraglutide (N=481) | Extension Period: Insulin Glargine (N=160)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Comparative Period: Insulin Glargine (N=484) | Comparative Period: Liraglutide (N=481) | Extension Period: Insulin Glargine (N=160)
Constipation (Gastrointestinal disorders) | 6 | 26 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 62 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 25 | 1
Nausea (Gastrointestinal disorders) | 13 | 146 | 2
Vomiting (Gastrointestinal disorders) | 8 | 46 | 1
Nasopharyngitis (Infections and infestations) | 38 | 35 | 12
Decreased appetite (Metabolism and nutrition disorders) | 1 | 45 | 0
Headache (Nervous system disorders) | 24 | 29 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any abstract/manuscript for comment at least 20/45 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.